CLINICAL TRIAL: NCT06441409
Title: Effect of Calorie-restricted Balanced Diet on Mobilization of Fat Storage Pools and Iron Deposition in Individuals With Obesity
Brief Title: Effect of Lifestyle Intervention on Mobilization of Fat Storage and Iron Deposition in Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22218; No. 2022JJ40749 (Other Grant/Funding Number: the Natural Science Foundation of Hunan Province)
Record Dates: First submitted 2024-04-15; First posted 2024-06-04 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-05

CONDITIONS: Liver Fat; Fertility Disorders; Life Style, Healthy; Glucose Metabolism Disorders (Including Diabetes Mellitus)
MeSH Terms: conditions — Fatty Liver; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Patients were intervened with lifestyle only.
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- lifestyle intervention (Experimental): Patients were intervened with lifestyle only and returned to clinic for tests in 6 months.
  Lifestyle intervention included the diet and exercise. Diet was an energy-restricted balanced diet. Exercise requires 5 days a week and 30 minutes every day.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Patients were intervened with lifestyle only and returned to clinic for tests in 6 months.
  Lifestyle intervention included the diet and exercise. Diet was an energy-restricted balanced diet. Exercise requires 5 days a week and 30 minutes every day.

SUMMARY:
The goal of this clinical trial is to learn if calorie-restricted balanced diet could uniquely influence various fat storage pools and iron deposition and explore the relationships between fat or iron deposition loss in specific locations and glucose metabolism. The main questions it aims to answer are:

After lifestyle intervention, which part of the body shows the fastest fat mobilization? Which part shows the slowest fat mobilization? Which area's fat mobilization is most related to the alleviation of glucose metabolism? Is there a relationship between the fat deposition in organs and the iron deposition in organs?

Researchers will compare the liver fat, pancreatic fat, visceral fat, subscutaneous fat, liver and pancrease iron depositon after lifestyle intervention using self pre-and post-control .

Participants will:

Receive the lifestyle intervention in outpatient. Visit the clinic once after 6 months for checkups and tests. Keep a diary of their diet.

DETAILED DESCRIPTION:
Fat mobilization status is assessed using magnetic resonance, while the relief of glucose metabolism is determined based on the results of the OGTT before and after life style intervention.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years
* have a BMI greater than 28.0 kg/m2
* exhibit abdominal obesity, defined as a waist circumference of at least 90 cm for men and 85 cm for women
* willing to undergo a 6-month lifestyle intervention

Exclusion Criteria:

* For newly diagnosed patients with type 2 diabetes: those with fasting blood glucose ≥ 11.1 mmol/L, random blood glucose ≥ 16.7 mmol/L, or HbA1c ≥ 9.0%, or those exhibiting significant hyperglycemic symptoms, who need to start antidiabetic medication treatment immediately;
* a prior history of pancreatic diseases;
* combination of drug-induced hepatitis, autoimmune hepatitis, and viral hepatitis;
* with a definitive diagnosis of diabetes who have already started medication treatment;
* severe complications from type 2 diabetes or other significant diseases;
* usage of drugs affecting body weight, insulin sensitivity, or metabolic-associated fatty liver disease in the past three months (such as insulin, glucocorticoids, thiazolidinediones, metformin, SGLT-2 inhibitors, or GLP-1 receptor agonists);
* with malignant tumors;
* acute or chronic infection;
* with elevated transaminase levels of unknown cause;
* hemochromatosis;
* with iron deficiency anemia who are receiving iron supplementation;
* who have donated blood or received a transfusion within the past six months;
* who have experienced cardiovascular events within the past six months;
* with acute or chronic blood loss;
* alcohol dependence, defined as ethanol intake exceeding 140 g/week for men and 70 g/week for women；
* pregnant and lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
The site-specific fat mobilization after 6 months' lifestyle intervention. | After 6 months intervention, patients were return to hospital for MRI analysis.
  Defined by percentage MRI-based fat loss. Calculated as (initial measurement minus follow-up measurement) / (initial measurement) × 100 and predefined to be assessed at 6-month follow-up. MRI scans were acquired with an INGENIA ELITION X (Philips Medical Systems Nederland B.V.).
The site-specific iron deposition mobilization after 6 months' lifestyle intervention. | Patients were return to hospital for MRI and serum tests after lifestyle intervention for 6 months.
  Defined by percentage MRI-based organ iron content loss. Calculated as (initial measurement minus follow-up measurement) / (initial measurement) × 100 and predefined to be assessed at 6-month follow-up. MRI scans were acquired with an INGENIA ELITION X (Philips Medical Systems Nederland B.V.).

SECONDARY OUTCOMES:
The correlation between liver fat and liver iron. | Patients were return to hospital for MRI and serum tests after lifestyle intervention for 6 months.
  Categorical variables were summarized as numbers (percentages), continuous variables with normal distributions as means (SDs), and continuous variables with non-normal distributions as medians (interquartile ranges [IQRs]). Treatment-induced changes were tested by the paired t test and Wilcoxon signed-rank test, as appropriate. The unpaired t test, Mann-Whitney U test, and Kruskal-Wallis test were used for group comparisons. Correlations between site-specific fat mobilization and clinical outcomes were investigated by calculating Pearson correlation coefficients and Pearson partial correlation coefficients. Two-sided P < 0.05 was considered statistically significant. Statistical analyses were performed using R software version 4.1.2 (http://www.r-project.org/).

CONTACTS AND LOCATIONS:
Overall Officials: Ping Jin, Study Chair — The Third Xiangya Hospital of Central South University
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hunan, China